CLINICAL TRIAL: NCT05977803
Title: Contribution of the CEST Sequence in the Characterization of Radionecrosis of Brain Metastases of Pulmonary Origin
Acronym: ACROP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP230263
Record Dates: First submitted 2023-06-21; First posted 2023-08-04 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Brain Metastases; Radionecrosis; Pulmonary Cancer
Keywords: radionecrosis, metastases,
MeSH Terms: conditions — Brain Neoplasms; Lung Neoplasms; Neoplasm Metastasis | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiation therapy (Other): Patient treated for metastatic cerebral lung cancer who has been treated with external beam radiotherapy such as in toto brain irradiation or stereotactic radiosurgery followed in the thoracic oncology department of Bichat Hospital.
  Interventions: Radiation: MRI with CEST sequence, IVIM and ASL sequence

INTERVENTIONS:
Radiation: MRI with CEST sequence, IVIM and ASL sequence — Three sequences will be added as part of the protocol (for an additional duration of about 10 minutes) :
  * The CEST sequence
  * The ASL infusion sequence
  * The IVIM sequence

SUMMARY:
The aim of the study is to determine whether the use of the CEST sequence would have diagnostic performance equivalent to the reference method of T2* infusion with contrast injection in the diagnosis of radionecrosis of lung cancer brain metastases.

DETAILED DESCRIPTION:
Brain metastases are frequent secondary sites in the evolution of cancers, with an incidence of all cancers combined of about 20% and up to 40% in the later phases of the disease. Among these metastases, the lung is the most common primary lesion (responsible for 20-56% of brain metastases). The overall prognosis for metastatic brain cancers is poor, with treatment-free survival of 1 to 2 months, and with treatment averaging 7-8 months. Their treatment is based on systemic medical treatment (chemotherapy, immunotherapy or targeted therapy depending on the status of the lesion) and on the other hand on the response to local treatment (surgery or radiotherapy). Radiotherapy is performed either as a first-line or post-operative depending on the resectability of the lesions and the operability of the patient.

Radionecrosis is a late complication (6 months to 2 years on average) and frequent (5-25%) of stereotactic radiotherapy. It may be promoted by the concomitant use of immunotherapy such as checkpoint inhibitors, which implies a probable increase in its incidence. Treatment of radionecrosis is based on corticosteroids; recent studies also propose Bevacizumab.

The distinction in MRI between tumor progression and radionecrosis is based on a multimodal approach. Indeed, conventional sequences alone have average performance (sensitivity 76% and specificity 59%). Several MRI methods have been evaluated, but their performance varies according to the studies. Cerebral perfusion is the most widely used method, requiring contrast injection with correct performance. However, there is no standardized perfusion value to directly extrapolate these results. MRI spectroscopy has also been studied, with correct performance but only evaluated on weak samples and retrospectively.

CEST is an MRI technique that uses endogenous contrast, i.e. does not require injection of contrast medium. It consists of specifically altering the signal of a molecular compound by causing saturation (i.e. cancellation of its signal) and studying the saturation of the solute (i.e. water) on contact. Indeed, due to a process called 'chemical saturation transfer', the signal from the water in contact with the targeted compound will also become partially saturated. The subtraction of the MRI signals acquired before and after saturation makes it possible to obtain a tissue mapping of the molecular compound initially targeted obtaining an indirect reflection of its concentration. Indeed, the macromolecular composition of tissues (inaccessible for physical reasons in spectroscopy) differs according to radionecrosis status or tumor progression, with more ""amide"" compounds in the second case.

This relatively recent development technique has been studied in primary and secondary brain tumors, especially in the context of radionecrosis, but mainly in primary brain tumors. It seems to allow a more precise and earlier detection of possible tumor progressions.

The diagnosis of radionecrosis is therefore a major step forward for the management of patients with irradiated brain metastases.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age
* Histologically proven primary lung cancer
* Histologically proven or not brain metastases
* Irradiated metastases
* Inclusion in a treatment protocol for brain metastases by brain metastasis in toto or stereotactic or gamma-knife radiotherapy
* Morphological increase of one or more lesions of secondary brain metastases on a follow-up MRI
* Patients affiliated to a social security scheme

Exclusion Criteria:

* Opposition to the study
* Contraindication to MRI
* Refusal of imaging by the patient
* Patient with state medical aid (unless exemption from affiliation)
* Severe cognitive impairment making informed consent impossible
* Patients under guardianship or deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Visually significant hyperperfusion on normalized cerebral blood flow mapping generated from T2* infusion data with injection, confirmed by quantitative measurement of a ratio > 2.5 between tumor DSC and contralateral white matter. | 24 months
  Diagnostic performance of the CEST sequence in the diagnosis of radionecrosis on irradiated metastases of primary lung cancer compared to injected T2* infusion sequence

SECONDARY OUTCOMES:
Diagnostic performances for the IVIM sequence using IVIM scattering derivatives: f', ADC | 24 months
Diagnostic performances for the ASL (arterial spin labeling) sequence using ASL infusion derivatives: intralesional CBF (cerebral blood flow) relative to contralateral white matter CBF | 24 months
Diagnostic performances of coupled CEST, IVIM and ASL sequences, evaluated by the derivates of the CEST sequence : APT-AUC (Area Under Curve), NOE-MTR (Magnetization Transfer Ratio) and NOE-AUC. | 24 months
Diagnostic performances of coupled CEST, IVIM and ASL sequences, evaluated by the derivates of the IVIM scattering : f', ADC | 24 months
Diagnostic performance of coupled CEST, IVIM and ASL sequences, evaluated by the derivates of the ASL infusion : intralesional CBF (cerebral blood flow) relative to contralateral white matter CBF | 24 months
Tolerance of acquisition of all CEST, IVIM and ASL sequences evaluated by the percentage of exams interrupted. | 24 months
Describtion of non-tumor white matter changes in the irradiation field and outside the CEST sequence irradiation field during follow-up | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Augustin Gaudemer, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Bichat-Claude Bernard, Paris, France